CLINICAL TRIAL: NCT01977534
Title: A Post-market Registry of Patients With de Novo Lesions in Previously Untreated Vessels Treated With Absorb BVS
Brief Title: To Study the Safety and Clinical Outcomes of the Absorb Bioresorbable Vascular Scaffold (BVS) System in Patients With de Novo Lesions in Previously Untreated Vessels
Acronym: ABSORB UK
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-304
Record Dates: First submitted 2013-10-18; First posted 2013-11-06 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: Bioabsorbable; Coronary Stent; Everolimus; drug eluting stents; stents; angioplasty; coronary artery disease; total coronary occlusion; coronary artery restenosis; stent thrombosis; vascular disease; myocardial ischemia; coronary artery stenosis; CAD; CAOD
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Absorb BVS: Subjects receiving Absorb BVS
  Interventions: Device: Absorb BVS

INTERVENTIONS:
Device: Absorb BVS — The Absorb BVS System is a bioresorbable poly(L-lactide) (PLLA) scaffold with a drug and bioresorbable polymer coating [formulation of everolimus in a bioresorbable poly(D,L-lactide) (PDLLA) coating].

SUMMARY:
The purpose of this study is to determine the safety and clinical outcomes of the Absorb BVS for daily use in patients with de novo lesions in previously untreated vessels.

DETAILED DESCRIPTION:
ABSORB UK registry is a prospective, single arm, post-market registry designed to:

* Provide ongoing post-market surveillance for documentation of safety and clinical outcomes of the Absorb Everolimus Eluting BVS System in daily percutaneous coronary intervention (PCI) practice per Instructions for Use (IFU, on-label use).
* Collect additional information (e.g. acute success) to evaluate handling and implantation of Absorb BVS by physicians under a wide range of commercial use conditions and following routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria must follow the most recent IFU which may include but are not limited to the following:

* Patient must be at least 18 years of age at the time of signing the Informed Consent Form
* Patient is to be treated for de novo lesions located in previously untreated vessels.
* Patient must agree to undergo all required follow-up visits and data collection.

Exclusion Criteria:

The exclusion criteria must follow the most recent IFU which may include but are not limited to the following:

* Inability to obtain a signed informed consent from potential patient.
* Patient belongs to a vulnerable population (per investigator's judgment, this also includes people with a direct link (hierarchical or financial benefit) to the registry Doctor or the registry Sponsor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the general interventional cardiology population
Sampling Method: Non-Probability Sample
Enrollment: 1005 (Actual)
Dates: Start 2014-01; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Acute Success: Device success (lesion based analysis) | From the start of index procedure to end of index procedure
  Achievement of a final in-scaffold residual diameter stenosis of < 50% assessed by online quantitative angiography or visual estimation, using Absorb BVS and without a device deficiency. A device is considered to have failed if it did not meet the requirements of the definition for clinical device success.
Acute Success: Procedural success (patient based analysis) | From the start of index procedure to end of index procedure
  Achievement of a final in-scaffold diameter stenosis of < 50% by online QCA or visual estimation using Absorb BVS, with or without any adjunctive devices, and without the occurrence of cardiac death, target vessel MI (Q-wave and non Q-wave MI), or repeat revascularization of the target lesion within 3 days of the index procedure.
Death (Cardiovascular, Non-Cardiovascular) | 1 year
Death (Cardiovascular, Non-Cardiovascular) | 3 year
Myocardial Infarction (MI) | 1 year
  Attributable to Q-wave MI (QMI), non-Q wave MI (NQMI), target vessel (TV), non-target vessel (NTV)
MI | 3 year
  Attributable to Q-wave MI (QMI), non-Q wave MI (NQMI), target vessel (TV), non-target vessel (NTV)
Target Lesion Revascularization (TLR) | 1 year
  all TLR
TLR | 3 year
  all TLR
TLR | 1 year
  clinically indicated (ID-TLR)
TLR | 3 year
  ID-TLR
Target Vessel Revascularization (TVR) | 1 year
  all TVR
TVR | 3 year
  all TVR
TVR | 1 year
  clinically indicated (ID-TVR)
TVR | 3 year
  ID-TVR
Cardiac Death/TV-MI/ID-TLR (Target Lesion Failure (TLF)) (Device-oriented endpoint) | 1 year
Cardiac Death/TV-MI/ID-TLR (Target Lesion Failure (TLF)) (Device-oriented endpoint) | 3 year
Cardiac Death/All MI/ID-TLR (MACE) | 1 year
Cardiac Death/All MI/ID-TLR (MACE) | 3 year
Cardiac Death/All MI/ID-TVR (Target Vessel Failure (TVF)) | 1 year
Cardiac Death/All MI/ID-TVR (Target Vessel Failure (TVF)) | 3 year
Scaffold/Stent Thrombosis | 1 year
  acute, sub-acute, late and very late
Scaffold/Stent Thrombosis | 1 year
  Definite, Probable
Scaffold/Stent Thrombosis | 3 year
  acute, sub-acute, late and very late
Scaffold/Stent Thrombosis | 3 year
  Definite, Probable

OTHER OUTCOMES:
Acute Procedural Analyses (all patients) | During the implantation procedure
  * Access site (femoral, brachial, radial)
  * Lesion preparation (Lesion 1, 2, 3, etc.)
    * Balloon pre-dilatation (yes - Max balloon size/Max balloon pressure, Cutting balloon yes/no, Other yes/no)
    * Techniques used to adequately prepare the lesion (de-calcification techniques (Rotablator yes/no, Other yes/no))
  * Treatment parameters
    * CASS numbers
    * No. of scaffolds per analyzable lesion (Lesion 1, 2, 3, etc.)
    * Scaffold length (Lesion 1, Lesion 2, Lesion 3, etc.)
    * Lesion length (Lesion 1, Lesion 2, Lesion 3, etc.)
    * Bailout / bailout device (if bailout required)
  * Post-treatment of lesion?
    * Balloon post-dilatation (no, yes - Max balloon diameter/Max balloon pressures/balloon length)
    * Jailed side-branch (no, yes). If yes, treatment of jailed sidebranch? (no, yes)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Baumbach, Principal Investigator — Bristol Heart Institute; Susan Veldhof, Study Director — Clinical Science
Locations (24):
- United Kingdom (24):
  - Lister Hospital, Stevenage, Hertfordshire
  - Basildon Hospital, Basildon
  - Royal Victoria Hospital, Belfast
  - Glan Clwyd District General Hospital, Bodelwyddan
  - Royal Bournmouth Hospital, Bournemouth
  - Sussex Cardiac Centre, Brighton
  - Bristol Heart Institute, Bristol
  - Papworth Hospital, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh
  - Frimley Park Hospital, Frimley
  - Golden Jubilee National Hospital, Glasgow
  - Leeds General Infirmary, Leeds
  - Glenfield Hospital, Leicester
  - Barts Heart Centre, London
  - Kings College Hospital, London
  - Northwick Park Hospital, London
  - Royal Brompton Hospital, London
  - Manchester Royal Infirmary, Manchester
  - James Cook University Hospital, Middlesbrough
  - The Freeman Hospital, Newcastle
  - Norfolk & Norwich University Hospital, Norwich
  - John Radcliffe Hospital, Oxford
  - Queen Alexandra Hospital, Portsmouth
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Baumbach A, Zaman A, West NEJ, O'Kane P, Egred M, Johnson T, Wheatcroft S, Bowles R, de Belder A, Bouras G, Lansky A, Hill J, Mathur A, de Belder MA, Banning AP. Acute and one-year clinical outcomes following implantation of bioresorbable vascular scaffolds: the ABSORB UK Registry. EuroIntervention. 2018 Jan 20;13(13):1554-1560. doi: 10.4244/EIJ-D-17-00886. PMID 29131802